CLINICAL TRIAL: NCT03844412
Title: Vestibulodynia: Understanding Pathophysiology and Determining Appropriate Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00100678; 1R01HD096331-01 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Vestibulodynia; Temporomandibular Disorder; Fibromyalgia Syndrome; Irritable Bowel Syndrome; Migraines; Tension Headache; Endometriosis; Interstitial Cystitis; Back Pain; Chronic Fatigue Syndrome
Keywords: Pelvic pain; Lidocaine; Estradiol; Nortriptyline; Chronic pain
MeSH Terms: conditions — Vulvodynia; Temporomandibular Joint Disorders; Fibromyalgia; Irritable Bowel Syndrome; Migraine Disorders; Tension-Type Headache; Endometriosis; Cystitis, Interstitial; Back Pain; Fatigue Syndrome, Chronic; Pelvic Pain; Chronic Pain | interventions — Nortriptyline

STUDY DESIGN:
Intervention Model Description: Two-center, randomized, double-blind, placebo-controlled 2x2 factorial study enrolling 400 women to participate for 24-week duration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- peripheral treatment (Active Comparator): 5% lidocaine/5 mg/ml 0.02% estradiol compound cream
  Interventions: Drug: 5% lidocaine/5 mg/ml 0.02% estradiol compound cream; Drug: Placebo pill
- central treatment (Active Comparator): tricyclic antidepressant nortriptyline pill
  Interventions: Drug: Nortriptyline; Drug: Placebo cream
- combined peripheral and central treatments (Active Comparator): 5% lidocaine/5 mg/ml 0.02% estradiol compound cream and tricyclic antidepressant nortriptyline pill
  Interventions: Drug: 5% lidocaine/5 mg/ml 0.02% estradiol compound cream; Drug: Nortriptyline
- placebo (Placebo Comparator): placebo cream and placebo pill
  Interventions: Drug: Placebo cream; Drug: Placebo pill

INTERVENTIONS:
Drug: 5% lidocaine/5 mg/ml 0.02% estradiol compound cream — Lidocaine/estradiol cream targets peripheral nerves and tissues affected in VBD. Participants will be provided with a diagram and written instructions, detailing how to apply the cream to the vaginal vestibule daily for weeks 1-16. Treatment with lidocaine/estradiol or placebo cream will be terminated at week 16 (end of month 4).
  Arms: combined peripheral and central treatments; peripheral treatment
Drug: Nortriptyline — Nortriptyline is a centrally-acting tricyclic antidepressant that is FDA-approved for treatment of neuropathic pain. Dosing will begin with one 10 mg pill nightly for week 1, then two 10 mg pills nightly for week 2, three 10 mg pills nightly for week 3, four 10 mg pills nightly for week 4, and five for weeks 5 -16. Treatment with nortriptyline or placebo pill will be tapered off over weeks 16-18, decreasing the dose by 10 mg every 4 days. Participants will be provided with a list of drugs to avoid that are known to interact with nortriptyline.
  Arms: central treatment; combined peripheral and central treatments
Drug: Placebo cream — The comparison treatment will be an identical-appearing placebo Moisturel™ cream
  Other Names: Moisturel cream
  Arms: central treatment; placebo
Drug: Placebo pill — The comparison treatment will be an identical-appearing placebo pill
  Arms: peripheral treatment; placebo

SUMMARY:
Vestibulodynia (VBD) is a complex chronic vulvar pain condition that impairs the psychological, physical, and sexual health of 1 in 6 reproductive aged women in the United States. Here, the investigators plan to conduct a randomized, double-blinded, placebo-controlled clinical trial to 1) compare the efficacy of peripheral (lidocaine/estradiol cream), centrally-targeted (nortriptyline), and combined treatments in alleviating pain and improving patient-reported outcomes and 2) determine cytokine and microRNA biomarkers that predict treatment response in women with distinct VBD subtypes. Positive findings from this study will readily translate to improved patient care, permitting the millions of women with VBD, their partners, and their clinicians to make more informed decisions about pain management.

DETAILED DESCRIPTION:
Vestibulodynia (VBD) is a chronic pelvic pain condition that affects 1 in 6 reproductive aged women, yet remains ineffectively treated by standard trial-and-error approaches. The investigators have identified two distinct VBD subtypes that may benefit from different types of treatment: 1) VBD peripheral (VBD-p) subtype characterized by localized pain specific to the vulvar vestibule, and 2) VBD central (VBD-c) subtype characterized by pain at both vaginal and remote body regions. Preliminary data further demonstrate that VBD-p and VBD-c subtypes differ with respect to patient reported outcomes (e.g., physical and mental health), production of cytokines (intracellular proteins that regulate the activity of pain nerves and inflammatory processes), and expression of microRNAs (small non-coding RNA molecules that regulate gene expression). Women with VBD-p exhibit normal psychological profiles; balanced circulating pro- and anti-inflammatory cytokines; and dysregulation in microRNAs that regulate the expression of genes in estrogen pathways. In contrast, women with VBD-c report decreased functional status and increased somatization; increased pro-inflammatory but not anti-inflammatory cytokines; and dysregulation in microRNAs that regulate the expression of genes relevant to muscle, nerve, and immune cell function. Based on these data, the investigators hypothesize that two VBD-p and VBD-c subtypes will preferentially respond to peripheral, central, or combined treatments and can be distinguished by cytokine and microRNA profiles. These hypotheses will be tested in a phase III clinical trial that evaluates diverse treatment strategies in women with VBD-p and VBD-c. Participants will be randomly assigned to one of four parallel arms: peripheral treatment with 5% lidocaine + 0.5 mg/ml 0.02% estradiol compound cream, 2) central treatment with the tricyclic antidepressant nortriptyline, 3) combined peripheral and central treatments, or 4) placebo. The treatment phase will last 4 months (with a 6-week titration at treatment initiation and 2-week taper period at 4 months), with outcome measures and biomarkers assessed at 4 time points (0, 2, 4, and 6 months). First, the investigators will compare the efficacy of treatments in alleviating pain among women with VBD-p and VBD-c using standardized tampon insertion with a numeric rating scale and self-reported pain on the McGill Pain Questionnaire. Next, the investigators will compare the efficacy of treatments in improving perceived physical, mental, and sexual health among women with VBD-p and VBD-c using standardized questionnaires. Finally, investigators will measure cytokines and microRNAs in women with VBD-p versus VBD-c using multiplex assays and RNA sequencing, and determine the ability of these biomarkers to predict treatment response. Successful completion of the proposed work will provide new insights into the mechanisms that drive pain perception and treatment response in two distinct VBD subtypes, and determine the efficacy of peripheral, central, and combined therapies in reversing this pain. Such findings will readily translate to improved patient care, permitting the millions of women with VBD, their partners, and clinicians to make more informed decisions about pain management.

ELIGIBILITY:
Inclusion Criteria

1. Female
2. Age 18-50 years
3. English-literate
4. Willingness to provide informed consent
5. Meeting criteria for diagnosis of VBD based on:

   1. self-report of 3 continuous months of insertional (entryway) dyspareunia, and/or pain to touch/tampon insertion
   2. pain score of ≥ 3 on the tampon insertion test

Exclusion Criteria

1. Use of daily topical lidocaine, or estradiol, or lidocaine/estradiol to the vulvar vestibule within the past three months
2. Use of nortriptyline or other TCA medications within the past three months
3. Use of pregabalin or gabapentin within the past three months
4. Presence of active dermatologic vulvar disease or vaginal infection
5. Untreated atrophic vaginitis (participants may undergo treatment and re-evaluation for enrollment if the condition is resolved)
6. Previous vestibulectomy
7. Pregnant or planning on becoming pregnant during the study period. Within the first six months of the postpartum period. Currently breastfeeding/lactating, or within three months of discontinuing breastfeeding/lactation.
8. Active incarceration
9. Cancer within the past year.
10. Chemotherapy and/or radiation treatment within the past year.
11. Unstable medical condition (e.g., renal impairment, significant hematological disease, cardiovascular disease, hepatic insufficiency, neurological disorder, autoimmune disease, or respiratory illness)
12. Clear inflammatory states (e.g., morbid obesity)
13. Use of immunosuppressant medications
14. History of intolerance to nortriptyline, topical lidocaine, or topical estradiol
15. Contraindications to use of nortriptyline: current use, or use within the past 3 months, of MAOIs, SSRIs, SNRIs, NDRIs; recent (within the past year) myocardial infarction, active psychotic or suicidal thoughts, narrow angle closure glaucoma
16. Contraindications to the use of lidocaine or local anesthetics
17. Contraindications to the use of topical estrogen therapy
18. Post-menopausal, defined as no menses for 12 consecutive months or surgical removal of both ovaries. (Hysterectomy is not an exclusion)
19. Have not had Botox of the pelvic floor muscles in the last 12 months, or pelvic nerve blocks in the last three months.
20. Are not currently enrolled or planning to enroll in another clinical trial during the course of this trial.
21. Are not currently receiving pelvic physical therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in pain score during the tampon test | Baseline, 16 weeks
  The Tampon Test will provide a self-reported numeric rating scale of pain with self-tampon insertion, performed by the patient and reported to the research nurse. Participants will be asked to verbally rate the pain on a scale of 0-10, with 0 meaning no pain and 10 meaning the worst possible pain.
Change in self-reported pain via the Short Form- McGill Pain Questionnaire (SF-MPQ) | Baseline, 16 weeks
  The SF-MPQ will be used to create a summary score. The SF-MPQ measures perceived sensory qualities of pain using 11 describers and affective qualities related to pain using 5 describers. Responses on 4-point scales are summed to compute scores for each section.
Change in self-reported physical/mental health via SF-12 Health Survey (SF12v2) | Baseline, 16 weeks
  The SF-12 assesses 6 domains: global health, physical functioning, physical roles, emotional functioning, emotional roles and pain interference using an algorithm based on answers to 12 physical and mental health-related questions.
Change in sexual health via Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 16 weeks
  The PROMIS score is based on a 96-item form developed by the NIH that measures 11 domains of biopsychosocial function and includes an assessment of sexual function measures (e.g., desire, frequency, fear, and pain) related to sexual intercourse.
Change in inflammation as measured by cytokine expression levels | Baseline, 16 weeks
  Cytokine expression levels will be measured via mesoscale discovery assays.
Change in regulators of pro-pain and pro-inflammatory genes, as measured by microRNA expression levels | Baseline, 16 weeks
  MicroRNA expression levels will be measured via sequencing read.

SECONDARY OUTCOMES:
Change in pain level as measured by Vaginal Vestibule Pressure Pain Intensities (PPI) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  Vaginal Vestibule PPIs will be determined using a cotton swab applied to 6 externally-accessed sites (at 12, 10, 7, 6, 5, 2 o'clock on the vestibule) for 1-2 seconds. Upon application of cotton swab at each site, participants will rate their pain intensity on a scale from 0-10.
Levator Muscle Complex Pressure Pain Thresholds (PPTs) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  Levator Muscle Complex PPTs will be determined using a digital vestibular algometer applied internally to the right, midline, and left puborectalis levator muscles sites (5, 6, and 7 o'clock) just lateral to the perineum.
Change in pain level as measured by Remote Bodily PPTs | Baseline, 8 weeks, 16 weeks, and 24 weeks
  Remote Bodily PPTs will be determined by applying the algometer to 3 'neutral' non-pelvic body sites (deltoid, shin, and trapezius), right and left, beginning at 1N and increasing until the participant's first sensation of pain. A composite score will be calculated.
Change in degree of overlapping pain, as measured by COPC follow-up survey | Baseline, 8 weeks, 16 weeks, and 24 weeks
  The COPC survey consists of 2 questions used to determine the change in degree of overlapping pain.
Change in mood as measured by the Symptom Checklist-27 (SCL-27) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  Symptom Check List 27 (SCL-27) questionnaire will be used to measure a broad range of psychological symptoms (e.g., anxiety and depression).
Change in somatic awareness via Pennebaker Index of Limbic Languidness (PILL) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  Pennebaker Index of Limbic Languidness (PILL) is used to create a summary score of somatic symptoms (e.g., itchy eyes, dizziness). Symptom frequency is recorded on a five-point Likert scale ranging from "never" to "more than once a week".
Change in perceived stress via Perceived Stress Scale (PSS) | Baseline, 8 weeks, 16 weeks, and 24 weeks
  The Perceived stress scale (PSS) is a 10-item scale that measures the impact of personal stress on thoughts and feelings.
Change in sleep as measured by the sleep scale | Baseline, 8 weeks, 16 weeks, and 24 weeks
  The sleep scale is a 12-item scale that measures amount of sleep and ease/difficulty of initiating and maintaining sleep.
Change in in pain score during the tampon test at other time points | 8 weeks and 24 weeks
  Change in pain score during the tampon test will be measured as described above.
Change in in pain score via the SF-MPQ at other time points | 8 weeks and 24 weeks
  Change in pain score via the SF-MPQ will be measured as described above.
Change in self-reported health on the SF12v2 at other time points | 8 weeks and 24 weeks
  Change in self-reported health on the SF12v2 will be measured as described above.
Change in self-reported health on the PROMIS at other time points | 8 weeks and 24 weeks
  Change in self-reported outcomes on the PROMIS will be measured. The PROMIS score is based on a 96-item form developed by the NIH that measures 11 domains of biopsychosocial function and includes an assessment of sexual function measures (e.g., desire, frequency, fear, and pain) related to sexual intercourse.
Change in cytokine biomarkers at other time points | 8 weeks and 24 weeks
  Change in cytokine levels will be measured as described above.
Change in microRNA biomarkers at other time points | 8 weeks and 24 weeks
  Change in microRNA levels will be measured as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Nackley, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data in a manner consistent with NIH's policy NOT-OD-14-124, found at http://grants.nih.gov/grants/guide/notice-files/NOT-OD-14-124.html, released August 28, 2014. Genotypic data (e.g. microRNA and protein expression) and relevant phenotypic data (e.g. pain scores) from 400 participants will be posted on the dbGaP website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The PI expects data release up to 6 months after data submission is initiated or at the time of acceptance of initial publication, whichever occurs first.
Access Criteria: Requests to download individual unit-record datasets should be submitted to the PI and require approval from a Data Access Committee convened by the NIH/NICHD.
URL: http://grants.nih.gov/grants/guide/notice-files/NOT-OD-14-124.html

REFERENCES:
- [Derived] Carey ET, Geller EJ, Rapkin A, Farb D, Cutting H, Akaninwor J, Stirling C, Bortsov A, McNulty S, Merrill P, Zakroysky P, DeLaRosa J, Luo S, Nackley AG. Rationale and design of a multicenter randomized clinical trial of vestibulodynia: understanding pathophysiology and determining appropriate treatments (vestibulodynia: UPDATe). Ann Med. 2022 Dec;54(1):2885-2897. doi: 10.1080/07853890.2022.2132531. PMID 36269028